CLINICAL TRIAL: NCT06259734
Title: Transfusion Camp for Medical Students in Rwanda: a Multidisciplinary Initiative Teaching Graduating Medical Students How to Utilize Blood Products and Derivatives Safely in District Hospitals
Brief Title: Transfusion Camp for Medical Students in Rwanda
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Rwanda (Other)
Responsible Party: Principal Investigator, Teresa Skelton, Clinical Assistant Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H23-04004
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Global Health; Medical Education

STUDY DESIGN:
Intervention Model Description: Data collection on the appropriateness of blood transfusion orders will be collected for educational course participants and compared with orders of physicians who did not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfusion Camp Rwanda course participants (Experimental): This group will participate in a 3 day course on best practices in Transfusion Medicine in Rwanda. They will participate in testing before and after the course to ascertain knowledge gained. They will then begin to work in hospitals ordering blood for their patients. Data collectors will access their blood product orders and determine the level of appropriateness of their orders based on the Rwanda Biomedical Centre National Transfusion Guidelines.
  Interventions: Behavioral: Transfusion Camp Rwanda education
- Intern Physicians not participating in Transfusion Camp (No Intervention): Blood product ordering practices with be assessed for appropriateness in physicians who did not participate in Transfusion Camp.

INTERVENTIONS:
Behavioral: Transfusion Camp Rwanda education — Transfusion Camp Rwanda 3 day education intervention covering all aspects of safe blood transfusion practices as per the Rwanda Biomedical Centre National Transfusion Guidelines
  Arms: Transfusion Camp Rwanda course participants

SUMMARY:
Transfusion medicine is closely linked with safe surgery. Transfusion Camp is a multidisciplinary educational project aimed at improving transfusion medicine knowledge in physicians. The course has been piloted in Rwanda, showing improvement in participant knowledge and confidence, resulting in its recommended implementation into the medical school curriculum.

This project aims to evaluate a multi-day Transfusion Camp course mandatory for graduating medical students and first-year interns practicing in district hospitals in Rwanda. Its implementation is evaluated through pre- and post-course testing, collecting participants' blood ordering practices following the course, and conducting participant interviews about barriers to safe transfusion medicine in their hospital.

DETAILED DESCRIPTION:
Purpose: to assess efficacy of the recommendation set out through the University of Rwanda faculty working group discussions and the Canada-Rwanda Transfusion Camp partnership to implement a mandatory, annual multi-day Transfusion Camp course for final year medical students preparing to enter internship training and dispersing across the majority of district hospitals in Rwanda.

Hypothesis: (1) Graduating medical students and new interns will have a statistically significant improvement in their test scores after a 3-day Transfusion Camp Rwanda course. (2) There will be a statistically significant positive change in blood product ordering practices among course participants when compared with interns who have not participated in Transfusion Camp Rwanda. (3) In conducting semi-structured interviews of participants who took part in Transfusion Camp Rwanda the investigators will identify key enablers and barriers that are faced by participants in patient blood management that will give insight on strategies for future research and interventions.

Population: Final year graduating University of Rwanda medical students about to enter their internship year at district hospitals in Rwanda and new interns currently in the first year of their internship at district hospitals in Rwanda.

Research method:

1. Knowledge assessment and course evaluation: A validated pre-test assessment used currently in Transfusion Camp Rwanda will be administered prior to and after the session is complete. This test is a regular component of all Transfusion Camp courses in Canada, the United Kingdom, and Rwanda and separate from the research component of this project. It is a portion of the standard Transfusion Camp curriculum.This assessment is a combination of knowledge-based multiple-choice questions, questions on confidence in carrying out transfusion medicine decision-making in patient care, and a brief course evaluation to inform future courses. After 3 months, a second post-test assessment will be administered in the same manner as the pre- and post-test to assess knowledge retention. This test also asks the question about whether or not participants have applied their new knowledge in clinical practice, which will give some insight into the applicability of the course work in Transfusion Camp to real-life transfusion problems in clinical practice in Rwanda.
2. Blood product ordering practices: blood ordering practices of intern physicians will be collected using the blood product order form currently in use at all laboratories and health centres in Rwanda for the ordering of blood products. Control data will be collected at district hospitals prior to Transfusion Camp: ordering practices of intern physicians at district hospitals who did not participate in Transfusion Camp and, where possible, the hospital does not have faculty who have previously participated in Transfusion Camp. Three months following Transfusion Camp, the blood ordering practices of Transfusion Camp participants will be collected over a three-month period.
3. Semi-structured interviews: Participants who indicated interest during Transfusion Camp will be contacted to consent to an interview three months post-Transfusion Camp to allow opportunity and time for the participants to apply what has been learned. The interviews aim to gain insight into contextual factors, including hospital culture, hierarchy, product availability, resources for continuing professional development, and anything else that may act as barriers to them being able to follow the Rwanda transfusion guidelines taught and reinforced in Transfusion Camp Rwanda. Interviews will preferably take place face-to-face with two interviewers, a Canadian faculty well experienced in the Transfusion Camp curriculum and one Rwandan faculty member who is also experienced in the curriculum but aware of the cultural context and able to communicate in Kinyarwanda as required.

ELIGIBILITY:
Inclusion Criteria:

* Final year graduating University of Rwanda medical students about to enter their internship year at district hospitals in Rwanda and new interns currently in their first year of their internship at district hospitals in Rwanda.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of appropriate transfusion orders | 3 months after Transfusion Camp Course
  The proportion of blood product transfusion orders classified as appropriate with 0 being no orders appropriate and 1 being all orders appropriate
Test score | End of 3 day course
  Mean change in test scores of course participants
Retention test score | 3 months after course
  Mean change in test scores of course participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
Only study investigators will have access to participant data. There is no plan to share this data beyond study investigators.